CLINICAL TRIAL: NCT03001245
Title: Interpersonal Counseling (IPC) for Treatment of Depression in Adolescents: Implementation and Effectiveness Study in School Health Care
Brief Title: Interpersonal Counseling (IPC) for Treatment of Depression in Adolescents
Acronym: IPCAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Collaborators: Ministry of Social Affairs and Health; Finland (Unknown); Finnish Institute for Health and Welfare (Other Government); City of Espoo (Unknown)
Responsible Party: Principal Investigator, Dr. Klaus Ranta, Head of Department, Department of Adolescent Psychiatry, Helsinki University Central Hospital, Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS 1277/2016
Record Dates: First submitted 2016-12-20; First posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Depressive Disorder
Keywords: adolescents; depression; psychotherapy; interpersonal therapy
MeSH Terms: conditions — Depressive Disorder; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPC (Experimental): Interpersonal Counseling
  Interventions: Behavioral: Interpersonal Counseling
- ST (Active Comparator): Standard treatment
  Interventions: Behavioral: Standard treatment

INTERVENTIONS:
Behavioral: Interpersonal Counseling — Interpersonal Counseling 1+6 sessions
  Arms: IPC
Behavioral: Standard treatment — Psychosocial treatment 1+6 sessions guided by the professional's standard professional principles and routinely available methods
  Arms: ST

SUMMARY:
The aim of this cluster randomized trial is to investigate whether the brief, 1+6 session psychosocial intervention, Interpersonal Counseling (IPC) is more effective than standard professional treatment (ST) in the treatment of mild or moderate depression among 12 to 17-year-old adolescents in services provided by school health care and counseling professionals (school nurses, school psychologists and school social workers). The clients are identified from the pool of adolescents routinely seen in school health care and counseling services.

A total of 54 school nurses, social workers, and psychologists from all public secondary schools in the standard education system of City of Espoo, Finland will be trained in IPC in a three-day workshop in two waves. Each school (plus the one primary care level health care unit for adolescents in Espoo) is represented by 1-3 trial IPC counselors. In the first wave the schools are cluster randomized to provide either A) 1+6 sessions of IPC, or B) 1+6 sessions of standard treatment (ST), which consists of psychosocial work as guided by the workers' own standard professional principles and methods. The workers randomized to deliver IPC get the IPC training immediately. In the second wave those who delivered ST in the first wave will be trained in IPC. The data for this trial will be collected from the first wave. The data collection period is one school year plus follow-up of clients after 3 and 6 months.

The clients are adolescents who have either self-referred themselves, are referred by other school personnel, or by parents to the services offered in the school due to emotional symptoms in the school year 2016 -2017 in the participating schools. They are screened with the BDI at the initial visit to identify depressive symptoms. A diagnostic interview will be administered to those exceeding a clinical cutoff. Main inclusion criterion is DSM-5 depressive disorder of either mild or moderate severity. Those with current harmful alcohol use, acute suicidal ideation or behavior, severe depression or anxiety disorder, psychotic symptoms or very low global level of functioning are excluded and offered other treatment.

The clients will complete self-report questionnaires (BDI) as outcome measures. Their level of depression symptoms will also be assessed with ADRS scale and their level of global psychosocial functioning with the CGAS by the project IPC counselors / ST providers. Moreover, the clients will complete the Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE) as a measure of global symptomatology after each session. A follow-up interview at 3 months and 6 months after treatment termination will be arranged. The K-SADS-PL will be used for diagnostic evaluation, the ADRS and the C-GAS to assess level of depressive symptoms and global functioning, and the adolescent completes both the BDI and YP-CORE as self-reports of symptomatology.

DETAILED DESCRIPTION:
Background:

The incidence of depression increases in adolescence. Depression is one of the most common and clinically mental health disorder in this age group. In total, 5-10 % of adolescents experience depression episodes, and among 1-2% of the age group depressive symptoms are persistent and long-term (Costello et al., 2011; Marttunen & Karlsson, 2010). Depression causes significant distress and functional impairment to those affected by it. Furthermore, depressions symptoms with onset in adolescents tend to predict symptom continuation or new episodes in adulthood, and they associate with increased risk of suicide, hospital treatment, psychosocial problems and concurrent anxiety, substance use, and conduct disorders (Weissman et al., 1999; Marttunen et al., 2015).

However, only a minority of adolescents with mental health disorders seek help. Possible reasons include lack of recognition of symptoms, stigma related to being referred to mental health services, and lack of expertise in treating hold mental health resources. Research also shows that intervening in the early phases of symptom expression is important (Horowitz & Garber, 2006) and that the longer the duration of a depressive episode is the poorer the outcome to even an evidence based treatment is (Curry et al., 2006). Thus, many factors support developing brief and effective interventions for treating mild/moderate depression in the immediate surroundings of adolescents, e.g. schools.

Interpersonal psychotherapy for adolescents (IPT-A; see Mufson, 2004a) is one of the evidence -based treatments for adolescent depression (Zhou et al., 2015). It is a 12-session treatment, which focuses in the interpersonal relationships of adolescents and their significance in relation to symptoms of depression. It has been shown to be effective in school-based mental health clinics (Mufson et al., 2004b). IPT-A is a 12-session treatment focusing on problems on one problematic area in interpersonal relationships (grief, interpersonal/role disputes, role transition, or interpersonal deficits/social isolation).

A short form of IPT, the one plus six-session interpersonal counseling (IPC) has been developed to address needs of depressive individuals in contexts where a brief intervention offers advantages (Weissmann et al., 2014). It has been shown to be effective when treating depressive symptoms of adults in primary level of care (Kontunen et al., 2015; Menchetti ym. 2014). IPC can be provided by healthcare workers and counseling personnel without mental health training (Weissman et al., 2014). IPC may also be suited especially well for adolescents with milder symptoms depression. Due to its brevity it may be especially suitable to be implemented in schools, where barriers formed by school curriculum and multiple tasks required of the school health care workers must be taken in account.

To date, few studies have investigated the efficacy and effectiveness of IPC in adolescent samples. Mufson et al. (2015) examined the feasibility of a brief, six-session version of IPT-A in a group of 12-19 in an open study finding support for its utility and feasibility in this age group. Currently, a pilot trial of IPC in an adolescent sample is ongoing in the UK (see: http://www.hra.nhs.uk/news/research-summaries/interpersonal-counseling-evaluation/). More data is needed about the feasibility of IPC among adolescents in school settings and its effectiveness as compared with routine care offered by school nurses, school social workers and school psychologists.

Aim: The purpose of this cluster randomized trial is to investigate whether the brief 1+6 session-long Interpersonal Counseling (IPC) is effective in the treatment of depressive symptoms among 13 to 16-year-old adolescents in the routine care provided by school health care professionals (consisting of school health care nurses, school psychologists and school social workers) who have been trained in IPC. The participants are adolescents who either seek help from these school heath care professionals or are referred to them by other school workers or their families.

Method:

Design, and training and supervision of the trial counselors:

The personnel working in school health care and counseling services from all of the 27 public upper secondary schools in the standard education system of the City of Espoo, and the personnel working in the only low-treshold primary level healthcare unit for adolescents in Espoo were invited to participate in the project as project IPC counselors. Altogether, 54 of them were willing to participate, i.e., to be trained in IPC and to deliver the treatment. The schools (and the one primary level clinic) were each represented by 1-3 workers.

After this, the schools (i.e. the workers working in each of them) were randomized to deliver either A) 1+6 sessions of IPC, or B) 1+6 sessions of standard treatment (ST), which consists of psychosocial intervention guided by the worker's routine professional's principles and standard work methods. The workers who were randomized to deliver IPC got the IPC training immediately. Those who were randomized to the ST group were instructed to deliver treatment by their normal professional standards and routine methods. The data collection period is one school year. After this time the participants in the RC group will be given IPC training.

The IPC training consists of one day basic training in IPT-A main principles plus two days of targeted IPC training by experienced experts in the field. The staff belonging to the arm who received IPC training (the project IPC counselors) are clinically supervised by clinicians working in secondary level psychiatry services who have both IPT-A and IPC training, throughout the data gathering period with the frequency of once in every two weeks.

Recruitment of clients:

The clients of this trial are adolescents who either self-refer themselves, are referred by other school personnel, or by their parents to the services offered in the school by school nurses, school social workers or school psychologists because of emotional symptoms in the school year 2016 -2017 in each of the participating schools. They are first screened on their first visit with a self-report instrument, the Beck Depression Inventory (BDI-21; Beck et al., 1961) to identify symptoms of depression. If they are present above the clinical cutoff for mild depressive symptoms, a clinical interview (K-SADS-PL adapted to DSM-5; see Kaufman et al., 1997) by a trained research coordinator follows. In this stage, the main inclusion criterion for the study, a diagnosis of a DSM-5 depressive disorder, severity either mild or moderate, is ascertained. As an exclusion criterion, current harmful alcohol use as assessed by AUDIT (Babor et al, 2001) is ruled out. Also the presence of acute suicidal ideation or behavior, severe depression or anxiety disorder, psychotic symptoms or very low global level of functioning are exclusion criteria, and if present these adolescents are offered other treatment. Those fulfilling the inclusion criteria are referred to either a project IPC counselor, or a project worker delivering ST, depending on the status of the school in the cluster randomization.

Interventions and measures:

IPC consists of one evaluation session, where symptoms of depression are reviewed and evaluated, and treatment is being offered, and six treatment sessions following the IPC protocol specified by Wilkinson et al. (personal notification). This manual is also used in a UK pilot trial of IPC for adolescents (see: http://www.hra.nhs.uk/news/research-summaries/interpersonal-counseling-evaluation/). It is compatible with Weissman's IPC manual (2014), and is developmentally tailored to reflect themes relevant to adolescents. Quite similarly, ST consists of one evaluative session, followed by six treatment sessions, which are guided by standard professional principles of the treating project worker and methods routinely used and available to her/him.

As primary outcome measures, the clients complete the BDI-21 (Beck et al., 1961) as a measure of the severity of depressive symptoms after first, fourth and sixth treatment session and the Young Person's Clinical Outcomes for Routine Evaluation (YP-CORE; Twigg et al., 2010) as a measure of global symptomatology after each session. As primary observer-rated outcome measures the project IPC counselor / project worker providing ST assess the severity of adolescent's depressive symptoms with the Adolescent Depression Rating Scale (ADRS, Revah-Levy ym. 2007) and the level of adolescent's global psychosocial functioning with the Child Global Assessment Scale (C-GAS; Shaffer et al., 1983) after first, fourth and sixth treatment session.

A follow-up interview after 3 months and 6 months after treatment termination is arranged. A research coordinator administers the K-SADS-PL (adapted for DSM-5, see Kaufman et al., 1997) the ADRS (Revah-Levy ym. 2007), the C-GAS (Shaffer et al., 1983) and the adolescent completes both the YP-CORE (Twigg et al., 2010) and the BDI-21 (Beck et al., 1961) questionnaires.

Statistical analysis:

We will use standard statistical methods for comparing IPC and RC groups. We will perform estimation of between-groups effect sizes between adolescent groups receiving IPC and ST on the primary outcome measures. A clinically significant change in the main outcome measure scores will be defined according to standard procedures. Given we also perform diagnostic evaluation at the onset of the treatment and at 3 months and 6 months follow-up, we estimate recovery and possible relapse in both groups.

Ethical considerations:

The Ethics Committee of Hospital District of Helsinki and Uusimaa has approved the study.

References Beck, A. T., Ward, C., & Mendelson, M. (1961). Beck depression inventory (BDI). Archives of General Psychiatry, 4, 561-71.

Costello, E. J., Copeland, W., Angold, A. (2011). Trends in psychopathology across the adolescent years: what changes when children become adolescents, and when adolescents become adults? Journal of Child Psychology and Psychiatry, 52, 1015-25.

Curry, J., Rohde, P., Simons, A., Silva, S., Vitiello, B., Kratochvil et al. (2006). Predictors and moderators of acute outcome in the Treatment for Adolescents with Depression Study (TADS). Journal of the American Academy of Child & Adolescent Psychiatry, 45, 1427-39.

Horowitz, L. J. & Garber, J. (2006). The Prevention of Depressive Symptoms in Children and Adolescents: A Meta-Analytic Review. Journal of Consulting and Clinical Psychology, 74, 401-15.

Kaufman, J., Birmaher, B., Brent, D., Rao, U., Flynn, C., Moreci, P. et al. (1997). Schedule for affective disorders and schizophrenia for school-age children - present and lifetime version (K-SADS-PL): Initial reliability and validity data. Journal of the American Academy of Child & Adolescent Psychiatry, 36, 980-88.

Kontunen, J., Timonen, M., Muotka, J. & Liukkonen, T. (2016). Is interpersonal counselling (IPC) sufficient treatment for depression in primary care patients? A pilot study comparing IPC and interpersonal psychotherapy (IPT). Journal of Affective Disorders, 189, 89-93.

Marttunen, M. & Karlsson, L. (2010). Course and treatment of adolescent major depression. Psychiatria Fennica, 41, 130-46.

Marttunen, M., Ranta K., Gergov, V., Strandholm, T., Ehrling, L., Tainio, V-M & Lindberg, N. (2015). Nuorten depression psykoterapeuttisten hoitomuotojen vaikuttavuus: Systemaattiseen hakuun perustuva kirjallisuuskatsaus. Suomen Lääkärilehti, 46, 3110-16. (Article in Finnish)

Menchetti, M., Rucci, P., Bortolotti, B., Bombi, A., Scocco, P., Kraemer, H. C., et al. (2014). Moderators of remission with interpersonal counselling or drug treatment in primary care patients with depression: randomised controlled trial. British Journal of Psychiatry, 204, 144-50.

Mufson, L., Dorta K. P., Moreau, D., Weissman, M. M. (2004a). Interpersonal psychotherapy for depressed adolescents. Guilford: New York.

Mufson, L., Pollack, D. K., Wickramaratne, P., Nomura, Y., Olfson, M., & Weissman, M. M. (2004b). A randomized effectiveness trial of interpersonal psychotherapy for depressed adolescents. Archives of General Psychiatry, 61,577-84

Mufson, L., Yanes-Lukin, P., & Anderson, G. (2015). A pilot study of brief IPT-A in primary care. General Hospital Psychiatry, 61,481-84

Revah-Lev, A., Birmaher, B., Gasquet, I., & Flissard, B. (2007). The Adolescent Depression Rating Scale (ADRS): a validation study. BMC Psychiatry, 7:2

Shaffer, D., Gould, M.S., Brasic, J. et al. (1983). A children's global assessment scale (CGAS). Archives of General Psychiatry, 40, 1228-31.

Twigg, E., Barkham, M., Bewick, B. M., Mulhern, B., Connell, J., & Cooper, M. (2010). The Young Person's CORE: Development of a brief outcome measure for young people. Counselling and Psychotherapy Research, 9, 160-68.

Weissman, M., Hankerson, S., Scorza, P., Olfson, M., Verdeli, H., Shea, S., et al. (2014). Interpersonal Counseling (IPC) for Depression in Primary Care. American Journal of Psychotherapy,68, 359-83.

Weissman, M. M., Wolk, S., Goldstein, R. B., Moreau, D., Adams, P., Greenwald, S., et al. (1999). Depressed adolescents grown up. JAMA, 281, 1707-13.

Zhou X, Hetrick SE, Cuijpers P, Qin B, Barth J, Whittington CJ et al. (2015). Comparative efficacy and acceptability of psychotherapies for depression in children and adolescents: a systematic review and network meta-analysis. World Psychiatry, 14, 207-22.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of DSM-5 Depressive Disorder (severity mild or moderate)

Exclusion Criteria:

* current harmful alcohol use
* acute suicidal ideation or behavior
* severe depressive disorder
* severe anxiety disorder
* psychotic symptoms
* very low global level of functioning

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Adolescent Depression Rating Scale after six scheduled treatment sessions | 6 weeks
Change from Baseline in Children's Global Assessment of Functioning after six scheduled treatment sessions | 6 weeks
Change from Baseline in Beck Depression Inventory after six scheduled treatment sessions | 6 weeks
Change from Baseline in Young Person's Clinical Outcomes for Routine Evaluation after six scheduled treatment sessions | one, two, three, four, five, and six weeks

SECONDARY OUTCOMES:
Change from Baseline in diagnostic status regarding depressive disorder assessed with Kiddie-Sads-Present and Lifetime Version 3 months after treatment termination | 3 months after treatment termination
Change from Baseline in diagnostic status regarding depressive disorder assessed with Kiddie-Sads-Present and Lifetime Version 6 months after treatment termination | 6 months after treatment termination
Change from Baseline in Adolescent Depression Rating Scale 3 months after treatment termination | 3 months after treatment termination
Change from Baseline in Adolescent Depression Rating Scale 6 months after treatment termination | 6 months after treatment termination
Change from Baseline in Beck Depression Inventory 3 months after treatment termination | 3 months after treatment termination
Change from Baseline in Beck Depression Inventory 6 months after treatment termination | 6 months after treatment termination
Change from Baseline in Children's Global Assessment Scale 3 months after treatment termination | 3 months after treatment termination
Change from Baseline in Children's Global Assessment Scale 6 months after treatment termination | 6 months after treatment termination
Change from Baseline in Young Person's Clinical Outcomes for Routine Evaluation 3 months after treatment termination | 3 months after treatment termination
Change from Baseline in Young Person's Clinical Outcomes for Routine Evaluation 6 months after treatment termination | 6 months after treatment termination

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Y Ranta, M.D., Ph.D., Study Chair — Hospital District of Helsinki and Uusimaa, Helsinki University Central Hospital; Mauri Marttunen, M.D., Ph.D., Study Director — University of Helsinki, Department of Adolesecent Psychiatry
Locations (1):
- Department of Adolescent Psychiatry, Helsinki University Central Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided